CLINICAL TRIAL: NCT00602173
Title: A Single Dose, Randomized, Three-Period, Three-Treatment, Crossover Bioequivalency Study of Cilostazol 100 mg Tablets Under Fasting Conditions
Brief Title: Bioequivalency Study of 100 mg Cilostazol Tablets Under Fasting Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Roxane Laboratories (Industry)
Responsible Party: Elizabeth Ernst, Director, Drug Regulatory Affairs and Medical Affairs, Roxane Labortories, Inc.
Organization: West-Ward Pharmaceutical (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CILO-03
Record Dates: First submitted 2008-01-15; First posted 2008-01-28 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Intermittent Claudication
MeSH Terms: conditions — Intermittent Claudication | interventions — Cilostazol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Cilostazol

SUMMARY:
The objective of this study was the bioequivalence of a Roxane Laboratories' Cilostazol Tablets, 100 mg, to PLETAL® Tablets, 100 mg (OTSUKA Pharmaceuticals) under fasting conditions using a single-dose, randomized, 3-treatment, 3-period, crossover design.

ELIGIBILITY:
Inclusion Criteria:

* No clinically significant abnormal findings on the physical examination, medical history, or clinical laboratory results during screening.

Exclusion Criteria:

* Positive test for HIV, Hepatitis B, or Hepatitis C.
* Treatment with known enzyme altering drugs.
* History of allergic or adverse response to Cilostazol or any comparable or similar product.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2003-05; Primary Completion 2003-05 (Actual); Study Completion 2003-05 (Actual)

PRIMARY OUTCOMES:
Bioequivalence | Baseline, Two period, Seven day washout

CONTACTS AND LOCATIONS:
Overall Officials: Daniel V Freeland, DO, Principal Investigator — CEDRA Clinical Research, LLC
Locations (1):
- CEDRA Clinical Research, LLC, Austin, Texas, United States